CLINICAL TRIAL: NCT03587129
Title: Clinical Study of Apatinib in the Treatment of Platinum Resistant Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient enter this study.
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201801
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer
Keywords: epithelial ovarian cancer; ovarian cancer; platinum-resistant; platinum-refractory
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): 1 times a day, atapinib, 500 mg, is taken orally
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — An anti-tumor Targeted drug
  Other Names: Apatinib mesylate

SUMMARY:
For patients with "Platinum-resistant recurrent ovarian cancer" after second-line chemotherapy failure Using apatinib as a single drug Clinical efficacy observation Single study no control

DETAILED DESCRIPTION:
The overall 5-year survival rate of ovarian cancer is 45%. The mortality rate of ovarian cancer accounts for the first in gynecologic cancer deaths. Ovarian cytoreductive surgery and postoperative platinum based chemotherapy are the standard treatment for advanced ovarian cancer. About 80% of ovarian cancer will eventually show relapse and metastasis. All patients with recurrent ovarian cancer will eventually develop into "platinum resistance". Platinum resistance was found in 1-6 months with platinum-free interval. There is no standard treatment protocol for recurrent ovarian cancer of "platinum resistant," usually with platinum-free single chemotherapy, such as: paclitaxel, docetaxel, liposomal doxorubicin, gemcitabine, topotecan and other. The response rate was 10%-30%, the median progression free survival was <4 months, and the median overall survival time was 12 months with platinum-free single-agent chemotherapy. The incidence of grade 3-4 hematologic or non-hematologic toxicity is about 40%. And chemotherapy has 14% mortality rate within 30 days of the start of single-agent chemotherapy in the literature reported. VEGF plays an important role in invasion and metastasis of ovarian cancer. VEGF directly stimulates tumor cell proliferation, growth and migration, and promotes ovarian cancer metastasis. The growth and metastasis of ovarian cancer cells are related to the quantity of VEGF. It has confirmed that inhibition of VEGF function can inhibit angiogenesis and inhibit the growth and metastasis of ovarian cancer cells in vivo experiments. The Chinese State Food and Drug Administration approved small molecular targeting drug, apatinib, for the treatment of advanced gastric cancer, for approval in December 13, 2014. The role of apatinib is the intracellular ATP binding site of VEGFR2 tyrosine receptor, which blocks the signal transduction of VEGF binding and leads to tumor angiogenesis inhibition. Apatinib can inhibit VEGFR2 effectively at a very low concentration, and a higher concentration can inhibit the platelet derived growth factor receptor (PDGFR), c-Kit and c-Src. Apatinib has only 20% grade 3-4 hematological and non hematological toxicity in the treatment of metastatic gastric cancer and gastro-esophageal junction adenocarcinoma. Deng et al reported one cases of progressive ovarian cancer. After 4-line chemotherapy resistance, a daily oral apatinib 500 mg was taken and a longer progression free survival (11.3 months) was obtained. Xie Congying et al of the First Affiliated Hospital of Wenzhou Medical University had a report in the 2017 ESMO conference. The report reviewed 15 cases of recurrent and metastatic ovarian cancer with a single drug atapatinib in the treatment of more than 2 lines of chemotherapeutic drug resistance. The median progression free survival was 5 months, the objective remission rate was 53.3% and the disease control rate was 73.3%. It is known from the above reports that apatinib has good efficacy and low toxicity in the treatment of "platinum resistant" recurrent ovarian cancer, but there is lack of prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years, signed informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. Patients must have a life expectancy of at least 3 months.
4. Histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary. Failure of at least two-line chemotherapy OR platinum resistant ovarian cancer (defined as relapsing within 6 months after a platinum based chemotherapy) OR platinum refractory ovarian cancer (defined as progressing during a platinum based chemotherapy).
5. Criteria for recurrence or metastasis: blood CA125 is more than 2 times the upper limit of normal value, or imaging findings (CT/MRI/PET-CT) show recurrence or metastasis, or ascites cancer cells are positive.
6. Platinum refractory or resistant criteria: relapse or metastasis within 6 months end of platinum based chemotherapy.
7. The interval time to last chemotherapy was more than 4 weeks.
8. The patient received radiotherapy or surgery for more than 4 weeks, and the wound healed completely.
9. Patients must have adequate organ function as defined by the following criteria: White blood cell count ≥ 3 x 10^9/L, Absolute neutrophil count (ANC) (≥ 1.0 x 10^9/L), Hemoglobin of ≥ 80 g/L, Platelets ≥ 70 x 10^9/L. Total bilirubin ≤ 1 x upper limit of normal (ULN), AST and ALT ≤ 2 x ULN. Serum creatinine ≤ 1 x ULN
10. The main organs (liver, kidney and heart) function are basically normal.

Exclusion Criteria:

1. Had prior exposure to apatinib or has known allegies to apatinib.
2. History of other malignant tumors (except those with cured basal cell carcinoma and cervical carcinoma in situ).
3. History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
4. Patients with QT interval prolongation.
5. Inadequately controlled hypertension.
6. Serious, non-healing wound, active ulcer, bowel obstruction.
7. History of abdominal fistula or gastrointestinal perforation within 28 days prior to Day 1.
8. Evidence of bleeding diathesis or coagulopathy.
9. Patients with positive urine protein.
10. Major surgical procedure within 28 days prior to Day 1.
11. Symptomatic central nervous system (CNS) metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Objective remission rate, ORR | 3 years
  Complete remission (CR) + partial remission (PR)

SECONDARY OUTCOMES:
progression- free survival, PFS | 3 years
  from entry time to disease progression or any cause of death
grade 3-4 hematologic or non hematologic toxicity | 3 years
  defined by CTCAE version 4.0
Overall survival | 3 years
  from entry time to death of any cause
disease control rate, DCR | 3 years
  Complete remission (CR) + partial remission (PR) + disease stability (SD)

CONTACTS AND LOCATIONS:
Overall Officials: ZhiPing Liu, MD, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
The investigators have no other clinical trial about ovarian cancer

REFERENCES:
- [Result] Parmar MK, Ledermann JA, Colombo N, du Bois A, Delaloye JF, Kristensen GB, Wheeler S, Swart AM, Qian W, Torri V, Floriani I, Jayson G, Lamont A, Trope C; ICON and AGO Collaborators. Paclitaxel plus platinum-based chemotherapy versus conventional platinum-based chemotherapy in women with relapsed ovarian cancer: the ICON4/AGO-OVAR-2.2 trial. Lancet. 2003 Jun 21;361(9375):2099-106. doi: 10.1016/s0140-6736(03)13718-x. PMID 12826431
- [Result] Alberts DS, Liu PY, Wilczynski SP, Clouser MC, Lopez AM, Michelin DP, Lanzotti VJ, Markman M; Southwest Oncology Group. Randomized trial of pegylated liposomal doxorubicin (PLD) plus carboplatin versus carboplatin in platinum-sensitive (PS) patients with recurrent epithelial ovarian or peritoneal carcinoma after failure of initial platinum-based chemotherapy (Southwest Oncology Group Protocol S0200). Gynecol Oncol. 2008 Jan;108(1):90-4. doi: 10.1016/j.ygyno.2007.08.075. Epub 2007 Oct 18. PMID 17949799
- [Result] Oronsky B, Ray CM, Spira AI, Trepel JB, Carter CA, Cottrill HM. A brief review of the management of platinum-resistant-platinum-refractory ovarian cancer. Med Oncol. 2017 Jun;34(6):103. doi: 10.1007/s12032-017-0960-z. Epub 2017 Apr 25. PMID 28444622
- [Result] Pujade-Lauraine E, Hilpert F, Weber B, Reuss A, Poveda A, Kristensen G, Sorio R, Vergote I, Witteveen P, Bamias A, Pereira D, Wimberger P, Oaknin A, Mirza MR, Follana P, Bollag D, Ray-Coquard I. Bevacizumab combined with chemotherapy for platinum-resistant recurrent ovarian cancer: The AURELIA open-label randomized phase III trial. J Clin Oncol. 2014 May 1;32(13):1302-8. doi: 10.1200/JCO.2013.51.4489. Epub 2014 Mar 17. PMID 24637997
- [Result] Rustin G, Vergote I, Micha JP, Duska LR, Reed N, Bendell J, Spitz D, Dark G, Hoch U, Tagliaferri M, Hannah AL, Garcia AA. A multicenter, open-label, expanded phase 2 study to evaluate the safety and efficacy of etirinotecan pegol, a polymer conjugate of irinotecan, in women with recurrent platinum-resistant or refractory ovarian cancer. Gynecol Oncol. 2017 Nov;147(2):276-282. doi: 10.1016/j.ygyno.2017.08.026. Epub 2017 Sep 19. PMID 28935273
- [Result] Roncolato FT, Joly F, O'Connell R, Lanceley A, Hilpert F, Buizen L, Okamoto A, Aotani E, Pignata S, Donnellan P, Oza A, Avall-Lundqvist E, Berek JS, Heitz F, Feeney A, Berton-Rigaud D, Stockler MR, King M, Friedlander M; GCIG Symptom Benefit group. Reducing Uncertainty: Predictors of Stopping Chemotherapy Early and Shortened Survival Time in Platinum Resistant/Refractory Ovarian Cancer-The GCIG Symptom Benefit Study. Oncologist. 2017 Sep;22(9):1117-1124. doi: 10.1634/theoncologist.2017-0047. Epub 2017 Jun 8. PMID 28596446
- [Result] Kaufman B, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmana J, Mitchell G, Fried G, Stemmer SM, Hubert A, Rosengarten O, Steiner M, Loman N, Bowen K, Fielding A, Domchek SM. Olaparib monotherapy in patients with advanced cancer and a germline BRCA1/2 mutation. J Clin Oncol. 2015 Jan 20;33(3):244-50. doi: 10.1200/JCO.2014.56.2728. Epub 2014 Nov 3. PMID 25366685
- [Result] Colombo N, Van Gorp T, Parma G, Amant F, Gatta G, Sessa C, Vergote I. Ovarian cancer. Crit Rev Oncol Hematol. 2006 Nov;60(2):159-79. doi: 10.1016/j.critrevonc.2006.03.004. Epub 2006 Oct 2. PMID 17018256
- [Result] Kyrgiou M, Salanti G, Pavlidis N, Paraskevaidis E, Ioannidis JP. Survival benefits with diverse chemotherapy regimens for ovarian cancer: meta-analysis of multiple treatments. J Natl Cancer Inst. 2006 Nov 15;98(22):1655-63. doi: 10.1093/jnci/djj443. PMID 17105988
- [Result] Webber K, Friedlander M. Chemotherapy for epithelial ovarian, fallopian tube and primary peritoneal cancer. Best Pract Res Clin Obstet Gynaecol. 2017 May;41:126-138. doi: 10.1016/j.bpobgyn.2016.11.004. Epub 2016 Nov 23. PMID 28027849
- [Result] Davis A, Tinker AV, Friedlander M. "Platinum resistant" ovarian cancer: what is it, who to treat and how to measure benefit? Gynecol Oncol. 2014 Jun;133(3):624-31. doi: 10.1016/j.ygyno.2014.02.038. Epub 2014 Mar 4. PMID 24607285
- [Result] Naora H, Montell DJ. Ovarian cancer metastasis: integrating insights from disparate model organisms. Nat Rev Cancer. 2005 May;5(5):355-66. doi: 10.1038/nrc1611. PMID 15864277
- [Result] Mu J, Abe Y, Tsutsui T, Yamamoto N, Tai XG, Niwa O, Tsujimura T, Sato B, Terano H, Fujiwara H, Hamaoka T. Inhibition of growth and metastasis of ovarian carcinoma by administering a drug capable of interfering with vascular endothelial growth factor activity. Jpn J Cancer Res. 1996 Sep;87(9):963-71. doi: 10.1111/j.1349-7006.1996.tb02127.x. PMID 8878460
- [Result] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Result] Deng L, Wang Y, Lu W, Liu Q, Wu J, Jin J. Apatinib treatment combined with chemotherapy for advanced epithelial ovarian cancer: a case report. Onco Targets Ther. 2017 Mar 13;10:1521-1525. doi: 10.2147/OTT.S126471. eCollection 2017. PMID 28352185
- See also: Surveillance, Epidemiology, and End Results program. — https://seer.cancer.gov/.